CLINICAL TRIAL: NCT06147856
Title: A Phase 1/2, First-in-Human, Open-Label, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of mRNA 3210 in Participants With Phenylketonuria
Brief Title: A Dose-finding Study to Evaluate mRNA-3210 in Participants With Phenylketonuria
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor no longer intends to recruit to this study.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3210-P101; 2023-506963-32-00 (Other: EU-CT Number)
Record Dates: First submitted 2023-11-18; First posted 2023-11-28 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Phenylketonuria
Keywords: mRNA-3210; Autosomal recessive genetic disorder; Central Nervous System Diseases; Nervous System Diseases; Brain Diseases; Metabolic Diseases; Phenylketonuria; In-born errors of metabolism; Phenylalanine; Rare metabolic disease
MeSH Terms: conditions — Phenylketonurias; Central Nervous System Diseases; Nervous System Diseases; Brain Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-3210 (Experimental): Participants will receive single dose of mRNA-3210 by intravenous (IV) infusion every 3 weeks (Q3W), every 2 weeks (Q2W), or every 1 week (Q1W) for up to 12 doses.
  Interventions: Drug: mRNA-3210

INTERVENTIONS:
Drug: mRNA-3210 — IV infusion

SUMMARY:
The main goal of this study is to assess the safety, and tolerability of multiple doses of mRNA-3210 in participants with phenylketonuria (PKU).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PKU due to phenylalanine hydroxylase (PAH) deficiency by molecular genetic testing from a central lab.
* At least 3 blood phenylalanine levels ≥600 micromole(μmol)/Litre (L) regardless of diet: 2 obtained during the screening period (at least 72 hours apart) and at least one historical value 6 to 24 months prior to start of screening.
* Have received documented approval from a study dietitian confirming that participant is willing and able to maintain dietary protein intake consistent with baseline intake during study participation.
* If applicable, maintained stable dose of neuropsychiatric medication (that is, for attention deficit hyperactivity disorder (ADHD), depression, anxiety, or other psychiatric disorders) prior to enrollment and willing to maintain stable dose throughout study participation unless, per investigator assessment, a change is clinically indicated.

Exclusion Criteria:

* Receipt of sapropterin or large-neutral amino acids within 14 days or 5 half-lives (whichever is longer) of the start of screening.
* Receipt of pegvaliase within 2 months of start of screening.
* For participants previously on pegvaliase: use or planned use of any injectable drugs containing polyethylene glycol (PEG), including medroxyprogesterone injection, within 3 months prior to the start of screening and during study participation with the exception of COVID-19 vaccinations.
* Receipt of any investigational drug within 30 days or 5-half-lives (whichever is longer) of screening.
* History of hypersensitivity to any component/excipient used in this study.
* Any other clinically significant medical condition that, in the Investigator's opinion, could interfere with the interpretation of study results or limit the participant's participation in the study

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2027-08-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Day 1 up to 52 weeks after EOT (up to 91 weeks)

SECONDARY OUTCOMES:
Change from Baseline in Blood Phenylalanine Levels | Day 1 up to 52 weeks after EOT (up to 91 weeks)
Maximum Observed Effect (Emax) | Day 1 up to 52 weeks after EOT (up to 91 weeks)
Area Under the Effect Versus Time Curve (AUEC) | Day 1 up to 52 weeks after EOT (up to 91 weeks)
Maximum Observed Concentration (Cmax) | Day 1 through Day 15 for Dose 1 and Dose 12
Area Under the Plasma Concentration-Time Curve (AUC) | Day 1 through Day 15 for Dose 1 and Dose 12
Number of Participants with Anti-Polyethylene Glycol Antibodies | Day 1 up to 52 weeks after EOT (up to 91 weeks)